CLINICAL TRIAL: NCT06047639
Title: Benefit of Bone Anchored Hearing Implants in Chronic Otitis Media
Brief Title: Bone Anchored Hearing Implants in Chronic Otitis Media
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Head of department of Otolaryngology, Pamukkale University
Other Study IDs: 14
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone Anchored Hearing Implants(BAHI) Patient: Patients with chronic otitis media whose hearing could not corrected with surgery and also could not use conventional and got bone-anchored hearing implants as a standard of care were included.
  Interventions: Device: Bone-anchored hearing implants

INTERVENTIONS:
Device: Bone-anchored hearing implants — surgically placed hearing device

SUMMARY:
The aim of this study is to investigate the cost, functional benefits, and impact on the quality of life of using bone-anchored hearing devices in chronic otitis media patients

DETAILED DESCRIPTION:
Hearing loss is a significant disability that disrupts an individual's communication with others and can have a profound impact on their social life and career. It can lead to social isolation, depression, anxiety, and even early dementia. Chronic otitis is one of the most important ear diseases that can cause hearing loss. Its treatment is surgical, but sometimes even after surgery, hearing rehabilitation is needed. In such cases, the first option is the use of hearing aids. Some patients may be unable to use hearing aids due to excessive ear canal clearance, recurrent ear infections, or outer ear canal problems. In such cases, bone-anchored hearing devices emerge as the most logical option, although they are more costly compared to regular hearing aids. The aim of this study is to investigate the cost, functional benefits, and impact on the quality of life of using bone-anchored hearing devices in the context of our country

ELIGIBILITY:
Inclusion Criteria:

* Adults
* No difficulty in coming to the hospital for follow-up
* Ability to communicate and express oneself at a level sufficient to interact with researchers
* Having an indication for BAHI due to Chronic Otitis media

Exclusion Criteria:

* Those with severe systemic illnesses (cancer, HIV, etc.)
* Psychiatric patients experiencing compliance issues with hearing tests
* Use of medication or medical devices that could affect the outcome of the study
* Patients who cannot adhere to regular follow-ups and do not use the device will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic otitis media whose hearing could not corrected with surgery and also could not use conventional and got bone-anchored hearing implants as a standard of care
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
free field hearing level | one year
  Measuring hearing threshold with device on
Speech, Spatial and Qualities of Hearing Scale | One year
  Subjective evaluation of the hearing by questionaries
World Health Organisation(WHO) Quality of Life Questionarie | One year
  Standard question list about the general health and quality of life of the patient

SECONDARY OUTCOMES:
Cost Benefit of the intervention | on year
  to calculate the health related expenses for the patient before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided